CLINICAL TRIAL: NCT02301754
Title: A First in Human Phase I Study of INVAC-1 as a Single Agent in Patients With Advanced Cancer
Brief Title: INVAC-1 Anti-Cancer hTERT DNA Immunotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invectys (Industry)
Collaborators: Keyrus Biopharma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INVAC1-CT-101
Record Dates: First submitted 2014-11-18; First posted 2014-11-26 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- INVAC-1 (Experimental): INVAC-1 at escalating doses of 100, 400 and 800 µg will be given as a single agent by intradermal injection (Q 4 weeks x 3 cycles), always combined with electroporation.
  Each patient will receive 3 cycles, unless motivated treatment interruption.
  Interventions: Biological: INVAC-1

INTERVENTIONS:
Biological: INVAC-1 — intradermal injection combined with electroporation

SUMMARY:
INVAC-1 is intended to be used for the treatment of adult patients with advanced solid tumors unresponsive to currently available therapies, or for whom no standard therapy is available.

DETAILED DESCRIPTION:
This is the first-in-patient study of INVAC-1, a DNA vaccine encoding human telomerase reverse transcriptase (hTERT). hTERT is the catalytic subunit of the telomerase complex which synthesizes telomeric DNA at the chromosome ends. hTERT is overexpressed in most human tumors and virtually all types of cancers.

INVAC-1 is developed for cancer therapy. Stimulation of the immune system directed against telomerase expressing cancer cells has the potential to generate tumor responses.

The study is designed to evaluate the safety and pharmacodynamics (PD) of INVAC-1 administered alone by intradermal route to adults with solid tumor malignancies.

As shown in non-clinical studies, the efficacy of the vaccine is enhanced by electroporation, which thus will be combined with the vaccination in the present study.

The general clinical plan includes development of INVAC-1 in both hematologic malignancies and solid tumors, as a single agent and in combination with other targeted anticancer agents such as check-points inhibitors, radiotherapy or chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of advanced/metastatic solid tumor malignancy
* Relapsed or refractory to standard treatment and for whom standard curative options do not exist
* Life-expectancy > 4 months
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* A delay of at least 3 weeks between last specific anticancer treatment and first INVAC-1 injection
* Adequate skin status
* Lack of biologically documented inflammation: C Reactive Protein < 15 mg/L
* No medical history of auto-immune disease
* Adequate bone marrow function
* Total white cells count ≤ 10 x 109/L (≤ 10,000/µL),
* Serum albuminemia > 30 g/L
* Adequate renal function, with an estimated creatinine clearance ≥ 50 mL/min as calculated using the Cockroft & Gault method
* Adequate liver function
* Adequate cardiac function
* Resolved acute effects of any prior therapy to baseline severity or Grade ≤ 1 CTCAE v. 4.03 except for Adverse Events not constituting a safety risk by investigator judgment
* Lack of immune-suppressive drugs and of high-dose corticoid treatment within 8 weeks prior to entering the study (prednisone or prednisolone ≤ 10 mg/day is allowed)
* Serum pregnancy test (for females of childbearing potential) negative within 7 days of first dose of study drug
* Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. Male patients must be surgically sterile or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator.
* Provision of written informed consent indicating that the patient has been informed of all the pertinent aspects of the trial to be followed
* Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

* Central Nervous System (CNS) primary or CNS metastatic malignancies
* Prior allogeneic hematopoietic stem cell transplant
* Chemotherapy, cancer immunosuppressive therapy, growth factors, systemic steroids, or investigational agents within 28 days before the first dose of study treatment
* Prior therapy with a compound of the same mechanism (immunomodulation) in the last 90 days prior to first dose of study drug
* Participation to a clinical trial of an experimental medication in the last 30 days prior to first dose of study drug
* Major surgery within 28 days of starting study treatment
* Radiation therapy within 28 days of starting study treatment
* Autoimmune disorders (eg, Crohn's Disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus) and other diseases that compromise or impair the immune system.
* Contra-indications to electroporation: cardiac pacemaker, any previous cardiac rhythm disorder, epilepsy.
* Active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness (HIV testing is not required).
* Unstable or serious concurrent medical conditions in the previous 12 months.
* Concurrent active malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix.
* Patients who are pregnant or breastfeeding.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality.
* Patients who are investigational site staff members or patients who are Invectys employees directly involved in the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11; Primary Completion 2018-02 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) of INVAC-1 as single agent in combination with electroporation | up to 28 days after last injection

SECONDARY OUTCOMES:
Adverse Events as characterized by type, frequency, severity (as graded by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v.4.03), timing, seriousness and relationship to study therapy INVAC-1 + electroporation; | up to 28 days after last injection
Routine laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v.4.03) and timing | up to 28 days after last injection
Tumor Necrosis Factor-α, Interleukine (IL)-17, IL-8, IL-6, IL-1β measured in serum | up to 28 days after last injection
anti-nuclear antibodies (ANA), anti-DNA, anti-TPO measured in serum | up to 28 days after last injection
Elispot Interferon gamma | every 4 weeks up to 3 months
Absolute cell counts and phenotype for circulating T and Natural Killer cells | every 2 weeks up to 3 months
circulating tumor DNA assessed by quantification of the allelic fraction of the DNA mutations; circulating DNA is extracted from plasma | before treatment; at day 15 of cycle 3
Objective response assessed by immune-related Response Criteria (ir-RC); | every 8 weeks during treatement and every 2 to 4 months during one-year follow-up
Duration of response | every 8 weeks during treatement and every 2 to 4 months during one-year follow-up
Progression free survival | approximately 15 months
Overall survival | approximately 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Culine, MD, Principal Investigator — Hopital St Louis - Paris - France
Locations (2):
- France (2):
  - Hôpital Saint Louis, Paris
  - Hôpital Européen Georges Pompidou, Paris

REFERENCES:
- [Derived] Teixeira L, Medioni J, Garibal J, Adotevi O, Doucet L, Durey MD, Ghrieb Z, Kiladjian JJ, Brizard M, Laheurte C, Wehbe M, Pliquet E, Escande M, Defrance R, Culine S, Oudard S, Wain-Hobson S, Doppler V, Huet T, Langlade-Demoyen P. A First-in-Human Phase I Study of INVAC-1, an Optimized Human Telomerase DNA Vaccine in Patients with Advanced Solid Tumors. Clin Cancer Res. 2020 Feb 1;26(3):588-597. doi: 10.1158/1078-0432.CCR-19-1614. Epub 2019 Sep 26. PMID 31558479